CLINICAL TRIAL: NCT02194920
Title: Arathyroid Reimplantation in Forearm Subcutaneous Tissue During Thyroidectomy: a Simple Way to Avoid Ipoparathyroidism and Evaluate Graft Function
Brief Title: Parathyroid Reimplantation in Forearm Subcutaneous Tissue During Thyroidectomy: a Simple Way to Avoid Ipoparathyroidism and Evaluate Graft Function
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe Cavallaro, Giuseppe Cavallaro, MD PhD, University of Roma La Sapienza
Other Study IDs: 06072011
Record Dates: First submitted 2014-07-03; First posted 2014-07-18 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Thyroid Goiter; Thyroid Carcinoma; Multinodular Goiter; Graves Diseases
MeSH Terms: conditions — Goiter; Thyroid Neoplasms | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Parathyroid reimplantation
  Interventions: Procedure: Thyroidectomy and parathyroid reimplantation in forearm subcutaneous tissue

INTERVENTIONS:
Procedure: Thyroidectomy and parathyroid reimplantation in forearm subcutaneous tissue

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of normal parathyroid tissue reimplantation in forearm subcutaneous tissue in case of accidental removal of parathyroid gland during thyroid surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by benign thyroid disease undergoing thyroidectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving thyroid surgery with accidental removal or devascularization of normal parathyroid gland
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Assessment of parathyroid tissue graft function by selective (left or right) parathormone measurement by vein blood sample | up to 3 months
  The primary outcome will be the assessment of reimplanted parathyroid function, evaluated by intact Parathormone (iPTH) measurement by separate blood samples (left and right arm) at 7 days, 1 month and 3 months after surgery. Ratio of 1.5 between the iPTH levels in the arm receiving graft and the opposite arm will be predictive of graft functionality

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Unit, ICOT Hospital, Latina, Italy